CLINICAL TRIAL: NCT01433692
Title: Does a BI Conducted by General Practitioners Reduce Consumption of Canabis in 15 to 25 Years Old ?
Brief Title: CANABIC : CANnabis and Adolescents, a Brief Intervention (BI) to Reduce Their Consumption
Acronym: CANABIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CHU-0103
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Addictions; Adolescents; Primary Health Care; Brief Intervention
Keywords: Addictions; Adolescents; Primary Health Care; Brief Intervention
MeSH Terms: conditions — Behavior, Addictive | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: Brief Intervention
- control group (Other)
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Brief Intervention — CANABIC is a quantitative study to validate use of BI with cannabis users: a randomized controlled trial, clustered study, comparing an intervention group (IG) and a control group (CG). The intervention is the achievement of the IB during a specific consultation. The outcome is the consumption of cannabic (Number of joints / month).

SUMMARY:
Background: Cannabis is the most prevalent illegal drug used in France, and consequences arising from the step of 'casual consumers'(1-10 joints/month). Side effects of cannabis are now well documented: Trauma (driving after consuming cannabis), respiratory, cardiovascular diseases and psychiatric and social problems. The general practitioner (GP) is the health professional most viewed by adolescents. Brief interventions (BI) for adult alcohol use have been shown to be efﬁcient. Some BI have been designed to inspect adolescents and consumption of cannabis have been piloted, showing their feasibility, but no test has validated them.

Aim : Does a BI conducted by general practitioners reduce consumption of canabis in 15 to 19 years old ?

Method:

Two preliminary qualitative studies (with adolescents and GP), were used to analyze the difficulties of communication around cannabis use. The Scientific Committee has analyzed the results and developed a workshop around BI, adapted to adolescents cannabis users.

CANABIC is a quantitative study to validate use of BI with cannabis users: a randomized controlled trial, clustered study, comparing an intervention group (IG) and a control group (CG). The intervention is the achievement of the IB during a specific consultation. The outcome is the consumption of cannabic (Number of joints / month).

The study will be carried out in 3 french regions : Auvergne, Rhône-Alpes and Languedoc-Roussillon. 150 GPs wil be recruited and randomized in intervention group or control group (ratio 1 :1).

Each GP will inlcude 5 adolescents (i.e. a total of 750 adolescents) - . The number of adolescents needed has been calculate with hypothesis of a significant difference of 30% in consumption of cannabis between adolescents who beneficied of BI (IG) and those who do not experienced BI ( CG) A pilot study has been conducted. Cannabis use by adolescents has decreased. Their perception of cannabis has changed: they are aware of the harmful effects of their consumption. This pilot study has improve many points of the protocol.

Results:

A decrease of 30% of consumption is expected (joints per month). Perception of cannabis by adolescents will be reviewed.

Conclusions:

To validate an IB adaptated to consultation with adolscents cannabis consumer in order to provide a tool for GP in their daily practice.

DETAILED DESCRIPTION:
General organisation of the study

* Recruitment of the GP: 3 months (from December 2011 to March 2012)
* Training of the intervention group GP during a one-day training, in March 2012, on 3 thematic: relationship between GP and adolescent, cannabis and BI; by an expert team
* Inclusion period : 10 months (from April 2012 to January 2013). The included patients will be followed for 12 months. There are 3 follow up consultations at 3, 6 and 12 months.
* First consultation used to the inclusion:

Information to the patient and collection of the patient non opposition (without informing the intervention objectives in the control group).

Evaluation of cannabis consumption, but also tobacco and alcohol consumption. Collection of the perception of cannabis by adolescents, and its impact on health.

Inclusion criteriae : repetead users : 1 to 10 per month; regular users : 11 to 29 per month; daily users : 1 and more per day.

In the IG : achievment of the BI with the adolescent. In each group, making appointment with the patient at 3 months

• Follow up consultations : At 3, 6 and 12 months. Evaluation of cannabis consumption, but also tobacco and alcohol consumption. Collection of the perception of cannabis by adolescents, and its impact on health.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 15 to 25 years Repetead users : 1 to 10 per month; regular users : 11 to 29 per month; daily users : 1 and more per day.

The patient must have given his informed consent and signed the form of no objection

Exclusion Criteria:

* Adolescents with psychiatric illness considered by the attending physician in acute decompensated
* Intellectual Disability
* Hard of hearing
* No French language skills
* Patient already under treatment for the withdrawal of an addicition to cannabis or other substance
* Adolescents who participated in the preliminary qualitative study

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
the number of joints consumed per month | at 12 months

SECONDARY OUTCOMES:
the number of joints consumed per month | at 3 and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine LAPORTE, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Laporte C, Lambert C, Pereira B, Blanc O, Authier N, Balayssac D, Brousse G, Vorilhon P. Cannabis users: Screen systematically, treat individually. A descriptive study of participants in a randomized trial in primary care. PLoS One. 2019 Dec 2;14(12):e0224867. doi: 10.1371/journal.pone.0224867. eCollection 2019. PMID 31790425
- [Derived] Laporte C, Vaillant-Roussel H, Pereira B, Blanc O, Eschalier B, Kinouani S, Brousse G, Llorca PM, Vorilhon P. Cannabis and Young Users-A Brief Intervention to Reduce Their Consumption (CANABIC): A Cluster Randomized Controlled Trial in Primary Care. Ann Fam Med. 2017 Mar;15(2):131-139. doi: 10.1370/afm.2003. PMID 28289112
- [Derived] Laporte C, Vaillant-Roussel H, Pereira B, Blanc O, Tanguy G, Frappe P, Costa D, Gaboreau Y, Badin M, Marty L, Clement G, Dubray C, Falissard B, Llorca PM, Vorilhon P. CANABIC: CANnabis and Adolescents: effect of a Brief Intervention on their Consumption--study protocol for a randomized controlled trial. Trials. 2014 Jan 30;15:40. doi: 10.1186/1745-6215-15-40. PMID 24479702